CLINICAL TRIAL: NCT03545412
Title: Clinical Study on the Application of a Non-Invasive Micro-Focused Ultrasound With Visualization System for Skin Laxity
Brief Title: Clinical Study on the Application of a Non-Invasive Micro-Focused Ultrasound With Visualization System for Skin Laxity (ULT-215)
Acronym: ULT-215
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULT-215
Record Dates: First submitted 2018-05-22; First posted 2018-06-04 (Actual); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-05

CONDITIONS: Facial Skin Laxity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microfocused ultrasound with visualization (Experimental)
  Interventions: Device: Microfocused ultrasound with visualization

INTERVENTIONS:
Device: Microfocused ultrasound with visualization — Each subject to receive a minimum of 800 treatment lines, on two planes of treatment using the 4-4.5mm and 7-3.0mm transducer depths
  Other Names: Ultherapy

SUMMARY:
To evaluate the effect of the Ulthera® system for facial laxity and sagging skin

ELIGIBILITY:
Inclusion Criteria:

1. Willing to sign a written consent form
2. Willing to have of facial skin laxity and wrinkles assessed by clinician
3. Male or female, aged 39 to 65 years.
4. Willingness to comply with protocol requirements, including returning for follow-up visits and abstaining from exclusionary procedures for the duration of the study.
5. Willingness to cooperate with photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
6. Must understand the ultrasound device (Ulthera) treatment may have no therapeutic effect.
7. Willingness and ability to provide written informed consent and HIPAA authorization prior to performance of any study-related procedure.

Exclusion Criteria:

1. Open wounds or lesions in the area(s) to be treated.
2. Severe or cystic acne on the area(s) to be treated.
3. Presence of an active systemic or local skin disease that may affect wound healing.
4. Active implants (e.g., pacemakers or defibrillators), or metallic implants in the treatment areas (dental implants not included.).
5. Subcutaneous fillers
6. Keloid scar
7. Patients with anticoagulant treatment plan.
8. Children, pregnant women, breastfeeding women.
9. Patients with the following disease conditions: bleeding disorders or coagulation disorder that may affect wound healing, active localized disease, herpes simplex, autoimmune diseases, diabetes, epilepsy bell-type paralysis (temporary facial palsy)

Ages: 39 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-01-10 (Actual); Primary Completion 2014-05-20 (Actual); Study Completion 2014-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lu PH, Yang CH, Chang YC. Quantitative Analysis of Face and Neck Skin Tightening by Microfocused Ultrasound With Visualization in Asians. Dermatol Surg. 2017 Nov;43(11):1332-1338. doi: 10.1097/DSS.0000000000001181. PMID 28945618

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 1 site in Taiwan.
Pre-assignment Details: A total of 25 participants were screened, enrolled and treated in the study.
Groups:
- Ultherapy Treatment: Participants received Ultherapy treatment to the facial areas including upper neck, cheek, brow, lateral orbit and infraorbital delivering a minimum of 800 treatment lines, on two planes of treatment using the 4-4.5 millimeter (mm) and 7-3.0 mm transducer depths.
Period: Overall Study
Arm/Group | Ultherapy Treatment
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all participants that were enrolled and treated with Ultherapy.
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 0
  African American/ Black | 0
  Hispanic/ Latino | 0
  Asian | 25
  Native Amer. Indian/ Alaskan Native | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 25
Body Mass Index (BMI) [Mean (Full Range); unit: kilogram per square meter (kg/m^2)] | 22.0 [18.6 to 26.0]
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Skin type I = white; very fair, red or blonde hair blue eyes; freckles; always burns, never tans, skin type II = white, fair, red or blond hair; blue, hazel or green eyes; usually burns, tans with difficulty, skin type III = cream white; fair with any eye or hair color (common); sometimes mild burn, gradually tans, skin type IV = brown; typical Mediterranean Caucasian skin; rarely burns, tans with ease, skin type V = dark brown; mid-eastern skin types; very rarely burns, tans easily, and skin type VI = black; never burns, tans very easily
  Participants
    Skin Type I | 0
    Skin Type II | 0
    Skin Type III | 3
    Skin Type IV | 22
    Skin Type V | 0
    Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improvement in Skin Laxity in Submental Region and Neck at Day 90
Description: Lift improvement as measured by quantitative analysis was considered greater than or equal to (>=) 20.0 square millimeter (mm^2) of the submental area Day 90 photograph compared to baseline photograph. The quantitative analysis was calculated by using five evenly spaced points on the neck. Area was calculated in between each of the 5 points and then sum of the five calculations was the total area of the region of interest.
Time Frame: Baseline, Day 90
Population: All participants enrolled and treated with Ultherapy. Only participants categorized as good candidates for photographs were included in the analysis. Good candidates for photographs was defined as those participants who had sufficient distance between the menton and neck, and enough lower face volume to allow for accurate measurements.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 13
Participants | 8

2. Primary Outcome: Number of Participants With Lift in Brow Region at Day 90
Description: Lift improvement as measured by quantitative analysis was considered minimum 0.5 millimeter (mm) Day 90 photograph compared to baseline photograph. The quantitative analysis was calculated by using five evenly spaced points along the natural outline of each participant's brow. Brow height was calculated using the sum and average of the five calculations in each brow area.
Time Frame: Baseline, Day 90
Population: All participants who were treated with Ultherapy were included for the assessment. The analysis included all participants who had the measurement available for brows. One participant excluded due to inability to measure brow.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 24
Participants | 12

3. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by the Principal Investigator Using the Global Aesthetic Improvement Scale (PGAIS) at Day 90
Description: Overall aesthetic improvement was assessed by the principal investigator using global aesthetic improvement scale (GAIS). At 90 days post-treatment, each principal investigator completed a GAIS, known as physician global aesthetic improvement scale (PGAIS) .The GAIS is 5-point scale (1-5), where: 1(very much improved); 2 (much improved); 3 (improved); 4 (no change); 5 (worse). Only participants who had any improvement were reported.
Time Frame: Baseline, Day 90
Population: All participants who were treated with Ultherapy were included for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 25
Participants | 21

4. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by the Subject Global Aesthetic Improvement Scale (SGAIS) at Day 90
Description: Overall aesthetic improvement was assessed by participants using global aesthetic improvement scale (GAIS). At 90 days post-treatment, each participant completed a GAIS, known as SGAIS.The GAIS is 5-point scale (1-5), where: 1(very much improved); 2 (much improved); 3 (improved); 4 (no change); 5 (worse). Only participants who had any improvement were reported.
Time Frame: Baseline, Day 90
Population: All participants who were treated with Ultherapy were included for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 25
Participants | 21

5. Secondary Outcome: Number of Participants With Improvement in Patient Satisfaction Questionnaire at Day 90
Description: Participants completed a PSQ at the 90-day visit. The PSQ has 5 satisfaction categories ranging from 'very dissatisfied' to 'very satisfied'.
Time Frame: Day 90
Population: All participants who were treated with Ultherapy were included for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 25
Participants | 21

6. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by the Physician Global Aesthetic Improvement Scale (PGAIS) at Day 180
Description: Overall aesthetic improvement was assessed by the principal investigator using the GAIS. At 180 days post-treatment, each principal investigator completed a GAIS, known as PGAIS .The GAIS is 5-point scale (1-5), where: 1(very much improved); 2 (much improved); 3 (improved); 4 (no change); 5 (worse). Only participants who had any improvement were reported.
Time Frame: Baseline, Day 180
Population: All participants who were treated with Ultherapy were included for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 25
Participants | 22

7. Secondary Outcome: Number of Participants With Overall Aesthetic Improvement as Assessed by the SGAIS at Day 180
Description: Overall aesthetic improvement was assessed by participants using GAIS. At 180 days post-treatment, each participant completed a GAIS, known as SGAIS. The GAIS is 5-point scale (1-5), where: 1(very much improved); 2 (much improved); 3 (improved); 4 (no change); 5 (worse). Only participants who had any improvement were reported.
Time Frame: Baseline, Day 180
Population: All participants who were treated with Ultherapy were included for the assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Ultherapy Treatment
Number analyzed (Participants) | 25
Participants | 20

ADVERSE EVENTS:
Time Frame: Baseline up to Day 180
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit.
Arm/Group | Ultherapy Treatment
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 19/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultherapy Treatment (N=25)
Contusion (Injury, poisoning and procedural complications) | 17
Application site edema (General disorders) | 3
Application site tenderness (General disorders) | 3
Hypersensitivity (Immune system disorders) | 1
Application site burn (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No